CLINICAL TRIAL: NCT07148726
Title: EFFECTS OF PYRROLOQUINOLINE QUINONE (PQQ) SUPPLEMENTATION ON METABOLIC AND PHYSIOLOGICAL ADAPTATION AT REST AND DURING SUBMAXIMAL EXERCISE IN NON-ENDURANCE-TRAINED ATHLETES: A RANDOMIZED PLACEBO-CONTROLLED TRIAL
Brief Title: EFFECTS OF PYRROLOQUINOLINE QUINONE (PQQ) SUPPLEMENTATION ON NON-ENDURANCE TRAINED ATHLETES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HEC-DSB/05-21
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Mitochondrial Biogenesis; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PQQ GROUP (Experimental): PQQ supplemented participants will receive 20mg/PQQ die
  Interventions: Dietary Supplement: Pyrrole Quinoline Quinone (PQQ)
- PLACEBO GROUP (Placebo Comparator): participants will be given a placebo for 36 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Pyrrole Quinoline Quinone (PQQ) — Subjects will be provided with 84 capsules of the PQQ or the placebo supplement. Both supplements were in capsule form and identical in size, shape and color. The PQQ content per capsule was 10 mg. The indication was to take two capsules every evening for 6 weeks. The duration of the supplementation protocol was assessed based on a previous study (Hwang et al., 2020), while the dose was chosen according to EFSA recommendations (Turck et al., 2017).
  Arms: PQQ GROUP
Other: Placebo — Subjects were provided with 84 capsules of placebo. The indication will be to take two capsules every evening for 6 weeks.
  Arms: PLACEBO GROUP

SUMMARY:
The aim of this study was to investigate the effects of six weeks of PQQ supplementation in non-endurance-trained individuals on:

1. physiological and metabolic response during a FATmax-VO₂peak exercise test
2. resting energy expenditure, body composition and blood biomarkers (fasting glucose, lactate dehydrogenase (LDH), creatine phosphokinase (CPK) and C-reactive protein (CRP) levels)
3. blood and urine omics markers of oxidative metabolism 24 basketball players will be randomized to consume a supplement containing 20 mg/day of PQQ or placebo (PLA) during a six-week intervention. Subjects will be encouraged to maintain their usual diet and training schedule. Body composition will be assessed by dual-energy-x-ray-absorptiometry and bioimpedance analysis. Aerobic exercise performance will be evaluated through a graded exercise protocol (six 5-minutes steps followed by n 2-minutes steps until exhaustion; the initial workload was 60 watts and increased by 35 watts at the end of each step) performed on a cycle ergometer. Capillary blood lactate samples were collected at the end of each step. Blood and urine samples were also collected, and metabolomics analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: Participants aged between 18 and 40 years.
* 2) Body mass index (BMI): BMI within the range of 18-30 kg/m².
* 4) Physical activity: Regular engagement in non-endurance physical activities (3-4 times a week), with no participation in structured endurance training programs.

Exclusion Criteria:

* 1) chronic disease;
* 2) acute illness; and
* 3) use of dietary supplements, pharmacological agents, or adherence to a hypocaloric diet.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Fat oxidation during FATmax-VO₂peak exercise test using gas analyzer. | 6 weeks
  Participants perform a graded exercise test on an electronically braked bicycle ergometer. A modified FATmax protocol is employed. After a 10-min warm-up at 50 W, the test commenced at 60 W and the workload increased by 35 W every 5 min until the participant could no longer maintain a cadence ≥60 rpm. The volume of Oxygen uptake (VO₂) and carbon dioxide production (VCO₂) per minute were recorded via a breath-by-breath gas analyzer. The average V̇O2 and V̇CO2 is extracted over the final 2 min of each stage of the test to ensure steady-state values . FatAT and carbohydrate (CHO) CHO oxidation and energy expenditure are calculated via stoichiometric equations (Jeukendrup & Wallis, 2005) and appropriate energy equivalents, with the assumption that the urinary nitrogen excretion rate was negligible. Data are analyzed workload-matched

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided